

### **Study Protocol**

Study ID: RCT-FP-01

**Title:** Clinical impact of a digital home-based falls prevention program on elderly people – a randomized controlled trial

**Document Version: 1.3** 

**Date:** 11/14/2018

Sponsor: SWORD Health, SA

Funding: P2020 Program

Research and Technological Development: I&D Individual Projects
- SWORD Care Project

### **Revision History**

| Version | Date | Description | Author |
|---------|------------|--------------------------------|--------|
| 1.0 | 25/01/2018 | Original version in Portuguese | FDC |
| 1.1 | 16/04/2018 | Translation to English | JG |
| 1.2 | 18/04/2018 | Content revision | FDC |
| 1.3 | 14/11/2018 | Content revision | MM |

### **Principal Investigator**

### Fernando Emanuel Dias Correia

Rua de Sá da Bandeira, number 651 1<sup>st</sup> right 4000-437 Porto

Contact: 966557789

### **Sub-Investigators**

### Dr.ª Mariana de Magalhães Sant'Ana

Rua de Vila Nova 10171, 4100 4100-503 Porto

Contact: 918448194

### Dr.ª Sofia Pinheiro Torres

Rua de Vila Nova 10171, 4100 4100-503 Porto

Contacto: 226165380

### **Investigation Center**

### **USF Aldoar**

Rua de Vila Nova 10171, 4100 4100-503 Porto

Contact: 226165380

Version 1.3

1. Introduction

Falls are a serious healthcare problem worldwide<sup>1,2</sup> and the third biggest

cause of chronic disability<sup>1</sup>. It is also estimated that falls are responsible for

20 to 30% of all injuries and for 10 to 15% of all emergency department

episodes<sup>3</sup>.

In the elderly population, falls are a particularly serious problem. Annually, it

is estimated that 28 to 35% of individuals aged 65 or over suffer a fall<sup>4,5</sup>, and

this percentage goes up to 32 to 42% in individuals over 70.

Besides age, there are several other risk factors for falls, which have been

reviewed elsewhere<sup>6,7</sup>. The most important are: a) living alone; b) previous

history of falls; c) presence of other chronic conditions (heart disease, chronic

obstructive lung disease, ostheoarthritis); d) previous stroke; e) cognitive

deficits; f) low vision; g) low body mass index; h) osteoporosis; i) multi-

medication (>4 concomitant drugs); j) psychotropic drugs (in particular

benzodiazepines); k) diuretics and some antiarrithmic drugs; l) proprioceptive

deficits.

The consequences of falls in the elderly population are more severe than in

other age groups. This results in a greater percentage of fatal falls<sup>8,9</sup>, but also

in the percentage of hospital admissions related to falls, corresponding to

7% of all admissions and to 85% of all accident-related admisisons in this

population  $^{10}$ . Falls can also lead to insecurity  $^{11}$ , fear of falling  $^{12}$  and loss of

independence <sup>13</sup>, worsening the problem even further.


With the aging world population, the number of falls is expected to increase<sup>1</sup>.

Without preventive measures, this increase can reach 100% by 2030<sup>14</sup>. Falls

prevention can help the older population in maintaining its independence

and quality of life, while reducing healthcare costs at the same time. 15

Physical exercise programs are one of the most effective tools in reducing the

risk of falls in the elderly population, and their validity has been confirmed in

several studies and meta-analysis<sup>15-18</sup>. To maximize their efficacy, these

programs should be performed regularly, be progressive<sup>19</sup>, have multiple

components (postural exercises, balance exercises and strength/endurance

exercises)<sup>16,17</sup> and be capable of promoting long-term engagement<sup>20</sup>.

Despite good results demonstrated by these programs, the biggest

challenge is to motivate older individuals to exercise and to maintain an

active lifestyle <sup>22</sup>. To maximize patient motivation, several authors stress the

need for a tailored program prescribed by a healthcare professional<sup>23-25</sup>,

additionally stating that the involvement of these professionals is one of the

main motivating factors to this population <sup>26</sup> and that even general advice or

brief telefone contacts can increase motivation <sup>27</sup>.

Besides the importance of involving healthcare professionals, physical activity

programs for this population need to be entertaining and stimulating <sup>24</sup>. This

helps explain why digital systems have evolved so rapidly <sup>28</sup>, with exergames

attracting particular interest <sup>29</sup>. Indeed, several studies demonstrate that

exergames are a viable and safe solution 30,31 and that they are more

engaging than comon exercise prescriptions 32,33.


Additionally, there is evidence showing an increase on clinical benefits and a

stronger engagement with physical activity programs when older people use

biofeedback-associated tracking and activity control devices <sup>28,34,35</sup>. Moreover,

given their potential benefits at such a low cost, biofeedback systems are

becoming increasingly appealing <sup>34</sup>.

Over the last few years, SWORD Health has developed a novel biofeedback

system - SWORD Phoenix® - based on inertial motion trackers that digitize

motion and use this information to provide real-time audiovisual feedback on

performance. SWORD Phoenix® takes advantage of biofeedback principles

to increase the efficiency of exercise programs. Plus, it maximizes

engagement through clean and user-friendly interfaces and gamification

strategies. Furthermore, SWORD Phoenix® allows users to perform their

rehabilitation sessions independently at home, under remote monitoring

from the clinical teams. This way, SWORD Phoenix® smart and efficiently

responds to the needs previously identified.

Given the dimension of the problem of falls in the elderly population and the

urgent need for a viable and cost-effective solution for falls prevention,

SWORD Health has created an exercise program aimed at this problem, and

integrated it within SWORD Phoenix®.

2. Study Design

This study is a single-center, prospective, non-blind, parallel-group,

randomized controlled trial with an intervention and a control group.


3. Study Objective

The aim of this study is to evaluate the clinical impact of a home-based falls

prevention program using a new biofeedback system - SWORD Phoenix® -

on community-dwelling older adults with fall risk in comparison with standard

of care.

The hypothesis is that the home-based falls prevention program using the

SWORD Phoenix® system will lead to a lower risk of falling than standard

medical care.

4. Study Outcomes

4.1 Primary outcome

The primary outcome will be the change in fall risk between the baseline and

the final assessment, measured through the "Five Times Sit to Stand Test".

4.2 Secondary outcomes

The secondary outcomes will be:

a) The change in fall risk between the baseline and the final assessment,

measured by the "Berg Balance Test".

b) The change in fall risk between the baseline and the final assessment,

measured by the "Timed Up and Go" test.

c) The change in fear of falling, through the change on "Falls Efficacy

Scale" score between the baseline and the final assessment.

d) The percentage of participants with falls in the study population

during the intervention period.


e) The percentage of participants with falls resulting in hospital

admissions or emergency care visits, during the intervention period.

5. Sample Size Estimation

The sample size calculation was performed considering the variable chosen

as the primary outcome - Five Times Sit to Stand Time (5XSST) - in a

superiority scenario.

To characterize the behavior of the primary outcome, a falls risk screening

was performed in a representative sample of the population consisting of 40

community-dwelling older individuals (>65 years old), followed at the

Unidade de Saúde Familiar de Aldoar (USF Aldoar), who met the inclusion

and exclusion criteria of this study. In this population, the mean score in the

5XSST was 19.67 seconds, with a standard deviation of 4.25.

Due to the lack of published data on the Minimal Clinically Important

Difference (MCID) for the 5XSST, we considered the MDC95 (Minimal

Detectable Change at the 95% confidence interval) reported by Goldberg et

al. <sup>36</sup> in a population of community-dwelling elderly women.

Considering a statistical power of 80%, a significance level of 0.05 (two-

tailed) and a dropout rate of 5%, 100 patients would be required to detect a

difference of 2.5 points between the two groups (50 in each group).

An interim statistical analysis on the results of the study will be performed

upon reaching the 70% inclusion mark. If the superiority of the intervention

group is demonstrated at this point, patient inclusion may be terminated.


6. Inclusion Criteria

a) Patients aged over 65 years old

b) Ability to walk at least 20 meters, unaided or with unilateral support

c) Ability to understand motor complex commands

d) Mini-Mental State Examination (MMSE) score > 24 points

e) Functional independence for instrumental activities of daily living

f) Risk of recurrent falls, defined as 5xSST score > 15,00 seconds

7. Exclusion Criteria

a) Patients residing in nursing homes, daycare units or assisted-living

facilities

b) Aphasia, dementia or psychiatric comorbidity, significantly interfering

with communication or compliance with a home-based exercise

program

c) Severe visual our hearing, interfering with communication or with

compliance to a home-based exercise program

d) Cardiac, respiratory or other condition incompatible with at least 30

minutes of light to moderate physical activity

e) Osteoarticular conditions (e.g. severe osteoarthrosis), which prevent

the patient from complying with a home-based exercise program

f) Patients with neurologic conditions (e.g. stroke, multiple sclerosis,

Parkinson's disease)

g) Other medical complications, which prevent the patient from

complying with a home-based exercise program

h) Illiteracy


8. Methods for identifying and recruiting patients

In each research center, the candidates for the study will be identified

through routine screening of patient lists from primary care consultations.

Whenever a candidate is identified for the study, the participant will be

approached by the investigator, who will explain the study in detail. The

prospective candidate will be given the patient information document

(Annex 1 - Information to Participants) and sufficient time to consider

whether he wishes to participate in the study.

Subsequently, the prospective candidate will be given the opportunity to

clarify any doubts, after which the informed consent form (Annex 2-

Informed Consent) will be signed and dated in duplicate by the patient and

the investigator. Only then will the randomization and baseline assessments

be performed.

9. Patient allocation to study arms

Patients will be randomized in a 1:1 ratio between arms, with randomization

blocks of 4 patients. Randomization will be performed centrally by the

online principal investigator - FDC - through an randomizer

(www.randomizer.org) and communicated by telephone to the investigator

responsible for data acquisition only after patient enrollment.

10. Blinding

The nature of the study does not allow blinding of the patients regarding

study arms. However, participants will be blinded to the primary and


secondary outcomes being measured. In addition, patient assessment will be

performed by one investigator blinded for data collection, for the

intervention administration and for the study arm. Statistic analysis will be

performed by a biostatistician blinded for the study arm.

11. Patient assessment

Patients will be assessed before the beginning of the intervention (AO), and

then every four weeks - week 4 (A4), 8 (A8) and 12 (A12). A follow-up

assessment will also be performed 12 weeks after the end of the intervention

(A24).

The assessments will be performed in a window of five working days before

or after the day on which the assessement should take place.

11.1 Baseline Assessment (AO)

In this assessment will be collected the following information:

a) Gender

b) Date of Birth

c) Educational Level (years)

d) Known fall risk factors

a. History of falls in the last year

b. Living alone

c. Chronic disease

i. DM

ii. Cardiac disease

iii. Respiratory disease (CPD/COPD)

iv. Osteoarticular disease (osteoarthrosis and osteoporosis)


d. Concomitant Medication

i. Number of medications

ii. Use of benzodiazepines or other sedative medication

iii. Use of antiarrhytmics

iv. Use of diuretics

e. Body mass index

f. Visual acuity loss

A multi-dimentional characterization of the participants' functional status will

also be performed, through specific performance tests (Five Times Sit to

<u>Stand Test</u> and <u>Timed up and Go Test</u>), a balance test (<u>Berg Balance Scale</u>)

and a self-reported fear of falling scale (Short Falls Efficacy Scale-

International) - see Annex 3: assessment scales and application

instructions.

The **5XSST** <sup>37</sup> is a performance test that measures the strength and the lower

limb mobility, which has been validated by Buatois et al. as a reliable marker

of falls risk in elderly community-dweller population 38. The same

investigators reported a cutoff value of 15 seconds to distinguish between

individuals with and without risk of recurrent falls <sup>39</sup>. Although the Minimal

Clinically Important Change has not been published for this test, Goldberg et

al reported an MDC95 (Minimal Detectable Change at the 95% confidence

interval) of 2.5 seconds in a elderly community-dweller women population <sup>36</sup>.

This test was chosen as the primary outcome for its proven validity, simplicity

of application, existence of a well-defined cutoff value and a well-defined

MCD95.


The **TUG** is a performance test that assesses the mobility, balance and gait in

elderly individuals and was developed in 1991 based on "Get up and Go

Test" 40. A shorter time indicates better performance, usually using the cutoff

level of 13.5 seconds to identify individuals at risk of falling in the community

<sup>45</sup>. However, the cutoff value reported in the literature varies between 10 and

33 seconds 46,47. The TUG is a fall risk assessment tool recommended by

several international guidelines <sup>48</sup>. However, a recent systematic review has

shown that this test has limited utility in the prediction of falls in the elderly

population inserted in the community, and should not be used alone for this

purpose 41.

The Berg Balance Scale (BBS) 42 was developed to evaluate the static and

dynamic balance in three domains: sitting, standing and changing posture. It

is a scale composed of 14 items graded by an external observer on 5 levels

(from 0 to 4). Scale scores range from 0 to 56, with higher scores

representing a higher level of functionality. The validity of this scale in the

prediction of fall risk was confirmed by several studies, including a recent

meta-analysis 43. However, there is no consensus regarding the cutoff level

used in the published studies (from 29 to 52 points), and this meta-analysis

suggested a cutoff level between 45 and 49 points to distinguish individuals

at low risk from the rest 51. In the absence of consensus on cutoff level, we

chose not to use this scale as the primary outcome of the study.

The Falls Efficacy Scale- International (FES-I) 44 was developed in order to

systematize on a scale the fear of falling. It is a questionnaire of 16 items

filled by the user, evaluating from 1 to 4 the fear of falling during the


execution of a series of activities of daily living. It is a standardized and

comparable measure over time, which provides an additional dimension in

the characterization of participants. To maximize its practical applicability, a

shortened version of the **Short Falls Efficacy Scale- International: Short** 

FES-I was developed and validated with 7 items (instead of 16) 53. Delbaere

et al. 45 subsequently validated the cutoff levels for Short FES-I: low fear (7-8);

moderate fear (9-13) and high fear (14-28). A recent study also showed that

this scale has a good correlation with objective fall risk measures such as TUG

55.

11.2 Interim assessments (A4 and A8), final assessment (A12) and follow-

up assessment (A24)

These assessments will be performed by an investigator blinded to the

randomization arm and will consist of:

a) TUG

b) 5XSST

c) BBS

d) FES

12. Intervention

Participants in the control group will benefit from standard medical care

currently in place at the participating primary care facility.

Participants within the experimental group will perform a 12-week falls

prevention program through SWORD Phoenix®, under remote monitoring

from a physical therapist. Participants will be asked to perform sessions at


least 3 days per week. In case of non-compliance with this periodicity, patients will not be excluded from the study, but will not be considered in "per protocol" analysis. Notwithstanding, daily sessions will be recommended (although not mandatory).

The program will consist of the following exercises:

| Exercise | Sets | Repetitions | Notes |
|---|---|---|---|
| Strengthening exercises | | | |
| Sitting exercises | | | |
| Sitting knee extension | 1 | 20 | Increase difficulty using ankle weights |
| Sit to Stand | 1 | 12 | |
| Standing exercises | | | |
| Standing hip abduction | 1 | 20 reps | |
| Standing knee flexion | 1 | 20 reps | |
| Squats | 1 | 12 reps | |
| Forward lunge with hold | 1 | 10 reps | |
| | Bala | nce exercises | |
| Single-leg stance | 1 | 10 reps | Patient will earn 1 star for |
| Single-leg stance with hip abduction | 1 | 10 reps | each 5 seconds, up to 25 seconds |
| Walking exercises | | | |
| March on the same spot | 1 | 40 steps | |
| Multi-directional steps | 1 | 20 steps | |
| Square walking | 1 | 5 reps | |

The exact composition of each program will be tailored according to the participant's specific needs, as defined by the physical therapist, i.e., it is not mandatory that every participant performs all exercises listed above.

The difficulty of each exercise (number of repetitions, series, weight addition or withdrawal of support) will be adjusted by the physical therapist, according the participant's stage and evolution.


**Face-to-face visits** 

Each study participant allocated to the experimental group will receive an

initial visit from the physiotherapist, which will be responsible for his

monitorization during the program. In this visit, an initial assessment of the

user's needs will be perfromed to define a tailored program. Training on the

system's usage will be given, and the first session will be carried out in the

presence of the therapist, to ensure that the user can interact autonomously

with the system (or leastwise caregiver-aided).

From this visit onwards, the participant will be monitored remotely by the

physical therapist, without subsequent face-to-face sessions. In the 4th and

8th weeks, each participant will receive a visit from the physical therapist for

reassessment and adjustment of the program. There will be no face-to-face

sessions during these two visits.

A follow-up telephone call will take place every two weeks (weeks 2, 6, 10).

Finally, extra visits or telephone calls can also me made, if necessary, and

these will be registered on patient's file (date, reason, duration).

Table 2 summarizes the interventional steps of the program:


Table 2. Schedule of face-to-face visits and telephone calls

| Week | Face-to-face visits | Telephone calls |
|------|---------------------|-----------------|
| 0 | Х | |
| 2 | | X |
| 4 | X | |
| 6 | | Х |
| 8 | X | |
| 10 | | X |
| 12 | X | |

### 13. Safety and adverse events

Patient safety will be ensured during all the process. For patients in the experimental group, safety will be evaluated through pain and fatigue scores (graduated from 0 to 10), collected at the end of each session. These will be presented to the patient using the mobile App and will be available for remote monitoring by the physical therapist. In case of excessive pain or fatigue, patients will be contacted to ascertain the cause and readapt prescription. Patients will also be instructed to report any other adverse events to their physical therapist by phone.

In the control group, in addition to the interim assessments, patients will be instructed to report any adverse events to a study investigator and, for this purpose, a direct phone contact will be provided.


All adverse events will be recorded on the participant's file (start date,

resolution date - if applicable), resolution status and severity).

14. Statistic analysis

To assess differences in clinical and demographic variables of the patients

allocated to the two study groups, independent samples test or Mann-

Whitney U test will be used for quantitative variables. For qualitative

variables, Chi-squared test Fisher's exact test will be used.

Outcome analysis will be performed using a "per-protocol" analysis. Patients

with adherence less than 43% (corresponding to at least 3 weekly sessions)

will not be considered on the "per protocol" analysis.

The impact of the interventions in the primary and secondary outcomes will

be evaluated considering the change between baseline and week 12.

Differences between the two study groups will be assessed using

independent samples test or Mann-Whitney U test.

Since outcomes will be measured in several different times during the

program, a repeated measures analysis will also be performed, using a

3x2/4x2 ANOVA, with group as an independent factor and time as a within-

subjects factor.

15. Potential risks and benefits to participants

There are no invasive procedures involved in this protocol and no relevant

risks are foreseen in both groups.

Participants in the control group will continue to benefit from the standard


medical care currently in place at the participating center, and thus no

increased associatred risk is expected in this study. Conversely, direct clinical

benefit from the study is not expected as well. However, participants will be

contributing to the development and testing of an innovative tool that could

have a significant positive impact on the older population's quality of life.

Participants in the experimental group will perform a falls prevention

program through SWORD Phoenix®, under remote monitoring of a physical

therapist. The therapist will have access to patient performance data, as well

as pain and fatigue scores, as rated by the patient at the end of each session.

This allows the therapist to detect adverse events and to act promptly. In

addition, no adverse events resulting from the use of SWORD Phoenix® have

been reported so far. Thus, participants in the intervention group are not at

increased risk and may directly benefit from the intervention, by improving

their muscular strength and balance and, consequently, by reducing falls risk.

16. Data protection

Data collection for this study was authorized by the National Commission on

Data Protection, with the authorization number 5457/2018. Personal data

will only be accessible to authorized individuals in this study. Personal data

will not be entered into the database as part of this research. The clinical

data collected will only be linked to the patient by a unique study number

and will contain no personal identifiers. Informed consent will be obtained

from participants to collect and retain this data. The data that will be used

for analysis and dissemination for research purposes will be completely

anonymized.


17. Ethical issues

All participants will be provided with information about the purpose and

procedures of the study and must give written informed consent before

inclusion.

The study was approved by the relevant Ethics Committee - Comissão de

Ética da ARS Norte (Chair: Prof Doutor Pedro Hespanhol) and will be

conducted in accordance with the relevant guidelines and regulations.

18. Dissemination of results

The results of the study will be published in peer-reviewed scientific journals

and presented at relevant national and international meetings.

19. System Technical Specifications

SWORD Phoenix® is a CE- and FDA- certified class I medical device

composed of the following components:

Inertial motion trackers

These are small high-precision motion trackers that capture and digitize the

user's motion, which is then transmitted via Bluetooth to the Phoenix App.

The motion trackers are fixed to Velcro straps placed in specific body

positions. To assist in the correct placement of the motion trackers, both the

trackers and the matching straps are color-coded. In this study, the following

setup will be used:

Red tracker: over the sternal manubrium


Green trackers: on the lateral surface of the leg, approximately

midway between the trochanter and the lateral epicondyle

Blue trackers: on the upper third of the antero-medial surface of

the tibia

Phoenix App

The App guides the patient in each exercise session. Before each exercise,

the patient is presented with a real-life video and audio explanation of that

exercise. The execution interface is subsequently shown, featuring a simple

and intuitive interface indicating the movement to be performed, a repetition

counter and a star counter. Patients earn stars for every correct repetition,

which is defined as a movement starting at the baseline and reaching or

surpassing a movement threshold, without violating movement or posture

constraints. In case the patient violates a movement constraint, a message is

prompted, showing which movement error was performed, so that the

patient can correct the movement in the following attempts. At the end of

each session, the patient is presented with a summary of the number of

completed repetitions and stars, as well as with rewarding badges for his

main achievments.

**Phoenix Portal** 

The portal is a web-based platform that allows the clinical team to create new

patient profiles and create exercise sessions for each patient. To prescribe a

session the clinician needs to select the exercises, number of sets and

number of repetitions. When a patient performs a session, the results are

uploaded to the platform and available for review. Based on this information,


the clinical team can edit the parameters of each exercise according to patient performance and progress.

### References

- 1. World Health Organization. WHO Global Report on Falls Prevention in Older Age. Community Health (2007). doi:978 92 4 156353 6
- 2. Day, L. et al. A protocol for evidence-based targeting and evaluation of statewide strategies for preventing falls among community-dwelling older people in Victoria, Australia. *Inj. Prev.* **17**, 1–8 (2011).
- 3. Scuffham, P., Chaplin, S. & Legood, R. Incidence and costs of unintentional falls in older people in the United Kingdom. *J. Epidemiol. Community Heal.* **57**, 740–744 (2003).
- 4. Prudham, D. & Evans, J. G. Factors associated with falls in the elderly: A community study. *Age Ageing* **10**, 141–146 (1981).
- 5. Campbell, A. J., Reinken, J., Allan, B. C. & Martinez, G. S. Falls in old age: A study of frequency and related clinical factors. *Age Ageing* **10**, 264–270 (1981).
- 6. NARI (National Ageing and Research Institute). 'An analysis of research on preventing falls and falls injury in older people: Community, residential care and hospital settings' (2004 update). Aust. Gov. Dep. Heal. Ageing, Dep. Heal. Ageing, Inj. Prev. Sect. (2004).
- 7. Todd, C. & Skelton, D. What are the main risk factors for falls amongst older people and what are the most effective interventions to prevent these falls? *World Health* 28 (2004).
- 8. Nevitt, M. C., Cummings, S. R., Kidd, S. & Black, D. Risk Factors for Recurrent Nonsyncopal Falls: A Prospective Study. *JAMA J. Am. Med. Assoc.* **261**, 2663–2668 (1989).
- 9. Phelan, E. A., Mahoney, J. E., Voit, J. C. & Stevens, J. A. Assessment and Management of Fall Risk in Primary Care Settings. *Medical Clinics of North America* **99**, 281–293 (2015).
- 10. Scott V, Pearce M, P. C. *Seniors' falls in Canada*. (Division of Aging and Seniors; Public Health Agency of Canada, 2005).
- 11. Tinetti, M. E. & Williams, C. S. Falls, injuries due to falls, and the risk of admission to a nursing home. *N. Engl. J. Med.* **337**, 1279–84 (1997).
- 12. Tinetti, M. E. & Williams, C. S. The Effect of Falls and Fall Injuries on Functioning in Community-Dwelling Older Persons. *Journals Gerontol. Ser. A Biol. Sci. Med. Sci.* **53A**, M112–M119 (1998).
- 13. Vellas, B., Cayla, F., Bocquet, H., de Pemille, F. & Albarede, J. L. Prospective study of restriction of activity in old people after falls. *Age Ageing* **16**, 189–193 (1987).
- 14. Kannus, P., Palvanen, M., Niemi, S. & Parkkari, J. Alarming rise in the number and incidence of fall-induced cervical spine injuries among older adults. *J. Gerontol. A. Biol. Sci. Med. Sci.* **62**, 180–3 (2007).


- 15. Salkeld, G. et al. Quality of life related to fear of falling and hip fracture in older women: a time trade off study. *BMJ* **320**, 341–6 (2000).
- 16. Gillespie, L. D. et al. Interventions for preventing falls in older people living in the community. Cochrane database Syst. Rev. 9, CD007146 (2012).
- 17. El-Khoury, F., Cassou, B., Charles, M.-A. & Dargent-Molina, P. The effect of fall prevention exercise programmes on fall induced injuries in community dwelling older adults: systematic review and meta-analysis of randomised controlled trials. *BMJ* **347**, f6234 (2013).
- 18. Cameron, I. D. et al. Interventions for preventing falls in older people in nursing care facilities and hospitals. *Cochrane Database Syst. Rev.* CD005465 (2010). doi:10.1002/14651858.CD005465.pub2
- 19. Sherrington, C. et al. Effective exercise for the prevention of falls: A systematic review and meta-analysis. J. Am. Geriatr. Soc. **56**, 2234–2243 (2008).
- 20. Delbaere, K. et al. Evaluating the effectiveness of a home-based exercise programme delivered through a tablet computer for preventing falls in older community-dwelling people over 2 years: Study protocol for the Standing Tall randomised controlled trial. BMJ Open 5, (2015).
- 21. Robertson, M. C., Campbell, A. J., Gardner, M. M. & Devlin, N. Preventing injuries in older people by preventing falls: A meta-analysis of individual-level data. *J. Am. Geriatr. Soc.* **50**, 905–911 (2002).
- 22. Pyae, A. et al. Investigating the Finnish elderly people 's attitudes and motivation towards digital game based physical exercises. Finnish J. eHealth eWelfare 9, (2017).
- 23. Nelson, M. E. et al. Physical activity and public health in older adults: Recommendation from the American College of Sports Medicine and the American Heart Association. *Medicine and Science in Sports and Exercise* **39**, 1435–1445 (2007).
- 24. Devereux-Fitzgerald, A., Powell, R., Dewhurst, A. & French, D. P. The acceptability of physical activity interventions to older adults: A systematic review and meta-synthesis. *Soc. Sci. Med.* **158**, 14–23 (2016).
- 25. Franco, M. R. et al. Older people's perspectives on participation in physical activity: A systematic review and thematic synthesis of qualitative literature. *British Journal of Sports Medicine* **49**, 1268–1276 (2015).
- 26. Schutzer, K. A. & Graves, B. S. Barriers and motivations to exercise in older adults. *Preventive Medicine* **39**, 1056–1061 (2004).
- 27. Bennett, J. A. & Winters-Stone, K. Motivating older adults to exercise: What works? Age and Ageing **40**, 148–149 (2011).
- 28. Vaziri, D. D. et al. Exploring user experience and technology acceptance for a fall prevention system: results from a randomized clinical trial and a living lab. Eur. Rev. Aging Phys. Act. **13**, 1–9 (2016).
- 29. Hasselmann, V., Oesch, P., Fernandez-Luque, L. & Bachmann, S. Are exergames promoting mobility an attractive alternative to conventional self-regulated exercises for elderly people in a rehabilitation setting? Study protocol of a randomized controlled trial. *BMC Geriatr.* **15**, 1–9 (2015).
- 30. Skjæret, N. *et al.* Exercise and rehabilitation delivered through exergames in older adults: An integrative review of technologies, safety and efficacy. *Int. J. Med. Inform.* **85**, 1–16 (2016).
- 31. Karahan, A. Y. et al. Effects of exergames on balance, functional mobility, and quality of life of geriatrics versus home exercise programme: Randomized controlled study.


- Cent. Eur. J. Public Health 23, S14-S18 (2015).
- 32. Karahan, A. Y. et al. Effects of exergames on balance, functional mobility, and quality of life of geriatrics versus home exercise programme: Randomized controlled study. *Cent. Eur. J. Public Health* **23**, S14–S18 (2015).
- 33. Meekes, W. & Stanmore, E. K. Motivational determinants of exergame participation for older people in assisted living facilities: Mixed-methods study. *J. Med. Internet Res.* **19**, (2017).
- 34. Alhasan, H., Hood, V. & Mainwaring, F. The effect of visual biofeedback on balance in elderly population: A systematic review. *Clin. Interv. Aging* **12**, 487–497 (2017).
- 35. Zijlstra, A., Mancini, M., Chiari, L. & Zijlstra, W. Biofeedback for training balance and mobility tasks in older populations: A systematic review. *J. Neuroeng. Rehabil.* **7**, 58 (2010).
- 36. Goldberg, A., Chavis, M., Watkins, J. & Wilson, T. The five-times-sit-to-stand test: Validity, reliability and detectable change in older females. *Aging Clin. Exp. Res.* **24**, 339–344 (2012).
- 37. Bohannon, R. W. Reference Values for the Five-Repetition Sit-to-Stand Test: A Descriptive Meta-Analysis of Data from Elders. *Percept. Mot. Skills* **103**, 215–222 (2006).
- 38. Buatois, S. et al. Five times sit to stand test is a predictor of recurrent falls in healthy community-living subjects aged 65 and older. J. Am. Geriatr. Soc. **56**, 1575–1577 (2008).
- 39. Buatois, S. *et al.* A Simple Clinical Scale to Stratify Risk of Recurrent Falls in Community-Dwelling Adults Aged 65 Years and Older. *Phys. Ther.* **90**, 550–560 (2010).
- 40. Podsiadlo, D. & Richardson, S. The timed 'Up & Go': a test of basic functional mobility for frail elderly persons. *J. Am. Geriatr. Soc.* **39**, 142–148 (1991).
- 41. Barry, E., Galvin, R., Keogh, C., Horgan, F. & Fahey, T. Is the Timed Up and Go test a useful predictor of risk of falls in community dwelling older adults: A systematic review and meta- analysis. *BMC Geriatr.* **14**, (2014).
- 42. Berg, K. O., Wood-Dauphinee, S. L., Williams, J. I. & Maki, B. Measuring balance in the elderly: Validation of an instrument. in *Canadian Journal of Public Health* **83**, (1992).
- 43. Park, S. H. & Lee, Y. S. The Diagnostic Accuracy of the Berg Balance Scale in Predicting Falls. Western Journal of Nursing Research **39**, 1502–1525 (2017).
- 44. Yardley, L. et al. Development and initial validation of the Falls Efficacy Scale-International (FES-I). Age Ageing **34**, 614–619 (2005).
- 45. Delbaere, K. et al. The falls efficacy scale international (FES-I). A comprehensive longitudinal validation study. Age Ageing **39**, 210–216 (2010).
- 56. Spencer MP, and Folstein MF. The Mini-Mental State Examination. In: PA Keller and LG Ritt (Eds). Innovations in Clinical Practice: A Source Book. Vol 4. Sarasota, FL: Professional Resource Exchange, Inc., 307-308, 1985.


### **ANNEX 1**

**INFORMATION TO PARTICIPANTS** 




# CLINICAL IMPACT OF A DIGITAL HOME-BASED FALLS PREVENTION PROGRAM ON ELDERLY PEOPLE - A RANDOMIZED CONTROLLED TRIAL

PARTICIPANT INFORMATION


This leaflet is intended to inform you of a clinical trial that USF Aldoar

and SWORD Health are currently undertaking.

What is the purpose of the study?

This study aims to assess the clinical impact of a home-based falls prevention

program using a new technology named SWORD Phoenix® in people over

65 years in risk of falling, compared to standard medical care.

What is SWORD Phoenix?

SWORD Phoenix® is a system composed of motion trackers placed on the

trunk and on lower limbs through Velcro straps. These trackers digitize your

movements and send this information to a mobile App (on a tablet). This App

guides you through the exercise sessions and tells you whether you are

performing them properly or not, helping you to correct any errors.

The information is then uploaded to an internet platform, where the clinical

team can remotely analyze the sessions, introducing changes as needed.

Thus, you will have a clinical team monitoring you remotely.

Is this study for me?

This study is intended for people over the age of 65, living in the community,


and who are at risk of falling. This leaflet was delivered to you because you

are a potential candidate to participate in the study.

What happens next?

If you agree to participate, and you meet the study criteria after an initial

assessment, you will be assigned to one of two groups: an experimental

group or a control group.

Participants in the experimental group will perform a falls prevention

program through the SWORD Phoenix® system, under the remote

supervision of a physical therapist. This program will last 12 weeks, during

which you must perform at least 3 exercise sessions per week. Throughout

the program, the sessions will be adapted by the physiotherapist according

to the performance.

Participants in the control group will continue to benefit from health care

routinely provided at the USF Aldoar, which includes fall risk assessment,

optimization of medication and information on how to prevent falls.

Participants in this group will not do any specific fall prevention program.


What are the risks associated with participating in the study?

There are no risks associated with participation in any of the groups, as no

risks arising from the use of the SWORD Phoenix® system are known.

Am I required to participate? And what are the costs?

No. Participation in this study is entirely voluntary and does not entail any

financial burden.

What happens if I do not want to participate?

If you do not want to participate, this will not have any negative

consequences to you. In this case, you will continue having your usual follow-

up with your Primary Care Physician.

Who will have access to my data?

Identification data will only be known to the trial investigators and will not be

made public under any circumstances.

All data collected will solely and exclusively be used for the production of

scientific articles that will always be anonymous, guaranteeing privacy and

the protection of participants's personal data.


If you have further questions about the study, please contact your Physician

or the Study Investigators through the following contacts:

Dr Mariana Sant'Ana:

Dr Fernando Correia: 966557789


### **ANNEX 2**

**INFORMED CONSENT** 




## CLINICAL IMPACT OF A DIGITAL HOME-BASED FALLS PREVENTION PROGRAM ON ELDERLY PEOPLE – A RANDOMIZED CONTROLLED TRIAL

**INFORMED CONSENT** 




### Clinical impact of a digital home-based falls prevention program on elderly people – a randomized controlled trial

### Informed Consent

I declare that I have received verbal and written information about the study in which I was invited to participate.

I read and understood all the information that was transmitted to me and had the opportunity to put the doubts that I thought necessary, which have been clarified to me.

I also understand my right to withdraw this study at any time, without having to give any explanation and without suffering any reprisals.

I understand that the results of the study can be published in Scientific Journals and used in other investigations, without any breach of confidentiality. I hereby authorize the use of the data for these purposes.

For these reasons, I agree to participate voluntarily in this study.

| Name of participant: | |
|----------------------------|-----------|
| Signature of participant: | |
| | Date: / / |
| Name of investigator: | |
| Signature of investigator: | |
| | Date: / / |




ASSESSMENT SCALES AND APPLICATION INSTRUCTIONS


MMSE (Mini-Mental State Examination)

The MMSE measures cognitive ability and begins with the assessment of

spatial and temporal orientation, with a maximum of 10 points. Then, two

aspects of memory are tested.

The first consists of the immediate memory of three orally presented objects,

followed by a serie of seven intercalated tasks that evaluate attention,

concentration and calculation, preventing the user from memorizing the

three previously learned objects. In this section a maximum of 11 points can

be obtained.

The last section assesses aphasia, testing naming, repetition, perceiving a

three-step command, reading, writing, and copying a drawing. A maximum

of 9 points can be obtained for a maximum total of 30 points.

I. ORIENTATION

1) Ask for: the year, season, date, day, month. Then ask specifically for

parts omitted e.g. "Can you also tell me what season it is?". One point for

each correct.

2) Ask in turn, "Can you tell me the name of this department? (state,

country, town, hospital, floor.)

**II. REGISTRATION** 

Ask the patient if you may test his memory. Then say the names of 3

unrelated objects, clearly and slowly, about one second for each. After you

have said all 3, ask him to repeat them. This first repetition determines his

score (0-3) but keep saying them until he can repeat all 3, up to 6 trials. If he

does not eventually learn all 3, recall cannot be meaningfully tested.


**III. ATTENTION AND CALCULATION** 

Ask the patient to begin with 100 and count backward by 7. Stop after 5

subtractions (93, 86, 79, 72, 65). Score the total number of correct answers. If

the patient cannot or will not perform his task, ask him to spell the word

"world" backward. The score is the number of letters in correct order, e.g.,

dlrow=5, dlorw=3.

IV. RECALL

Ask the patient if he can recall the 3 words you previously asked him to

remember in the registration section. Score 0-3.

V. LANGUAGE

**NAMING:** Show the patient a wrist watch and ask him what it is. Repeat for

pencil. Score 0-2.

**REPETITION:** Ask the patient to repeat the sentence "No ifs, ands, or buts"

after you. Allow only one trial. Score 0-1.

**3 STAGE COMMAND**: Give the patient a piece of plain blank paper and ask

him to follow your instructions: "Take the paper in your right hand, fold it in

half and put it on the floor." Score 1 point for each part correctly performed.

**READING:** On a blank piece of paper, print the sentence, "Close your eyes,"

in letters large enough for the patient to see clearly. Ask him to read it and

do what it says. Score 1 point only if he actually closes his eyes.


WRITING: Give the patient a blank piece of paper and ask him to write a

sentence for you. Do not dictate a sentence. It is to be written

spontaneously. It must contain a subject and a verb and be sensible. Correct

grammar and punctuation are not necessary.

COPYING: On a clean piece of paper, draw two intersecting pentagons,

each side about 1 inch, and ask him to copy it exactly as it is. All 10 angles

must be present and 2 must intersect to score 1 point. Tremor and rotation

are ignored.


### Timed up and Go Test

The Timed Up and Go is a test that assesses mobility, balance, walking ability in older adults.

To perform the test, follow the instructions:

- 1) Select a chair with armrests and a seating height of 44-47 cm
- 2) Measure 3 meters in a straight line from the chair and place a mark on the floor
- 3) Ask the patient to sit in a chair with his/her back against the chair back
- 4) Instruct the patient to rise from the chair on the command "go", walk 3 meters at a comfortable and safe pace, turn, walk back to the chair and sit down
- 5) Begin timing at "go" and stop when the patient is seated
- 6) Register the time with two decimal digits in the patient file


**Five Times Sit to Stand Test** 

The Five Times Sit to Stand Test is a functional measure of lower limb

muscle strength that quantifies the functional change of transitional

movements.

To perform the test, follow the instructions:

1) Select a chair with armrests and ask the patient to sit in the middle

of the seat with arms crossed behind the neck or arms crossed with

hands touching the shoulders. Advise the patient to keep their feet

on the ground and correct posture

2) Instruct the patient to rise from the chair and sit five times as fast as

possible on the command "start"

3) Ask the patient to stand up completely between the test repetitions

and not touch the back of the chair during each repetition

4) The counting begins on the command "start" and ends when the

hips are in contact with the chair after the fifth repetition.

5) Register the time with two decimal digits in the patient file

(maximum 2 minutes)

6) Failure to complete the five repetitions without assistance or

support from the upper limb indicates non-compliance with the

test.


### **Berg Balance Scale**

### Description:

14-item scale designed to measure balance of the older adult in a clinical setting.

Equipment needed: Ruler, 2 standard chairs (one with arm rests, one without)
Footstool or step, Stopwatch or wristwatch, 15 ft walkway

### Completion:

Time:

15-20 minutes

Scoring:

A five-point ordinal scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Total Score = 56

Interpretation:

41-56 = low fall risk

21-40 = medium fall risk0-20 = high fall risk

### Criterion Validity:

"Authors support a cut off score of 45/56 for independent safe ambulation".

Riddle and Stratford, 1999, examined 45/56 cutoff validity and concluded:

- Sensitivity = 64% (Correctly predicts fallers)
- Specificity = 90% (Correctly predicts non-fallers)
- Riddle and Stratford encouraged a lower cut off score of 40/56 to assess fall risk

Comments: Potential ceiling effect with higher level patients. Scale does not include gait items

### Norms:

Lusardi, M.M. (2004). Functional Performance in Community Living Older Adults. Journal of Geriatric Physical Therapy, 26(3), 14-22.

Table 4. Berg Balance Scale Scores: Means, Standard Deviations, and Confidence Intervals by Age, Gender, and Use of Assistive Device

| Age (y) | Group | N | Mean | SD | CI |
|---------|-----------|-----|------|------|-------------|
| 60-69 | Male | -1. | 51.0 | - | 35.3 - 66.7 |
| | Female | 5 | 54.6 | 0.5 | 47.6 - 61.6 |
| | Overall | 6 | 54.0 | 1.5 | 52.4 - 55.6 |
| 70-79 | Male | 9 | 53.9 | 1.5 | 48.7 - 59.1 |
| | Female | 10 | 51.6 | 2,6 | 46.6 - 56.6 |
| | Overall | 19 | 52.7 | 2.4 | 51.5 - 53.8 |
| 80-89 | Male | 10 | 41.8 | 12.2 | 36.8 - 46.8 |
| | Female | 24 | 42.1 | 8.0 | 38.9 - 45.3 |
| | No Device | 24 | 46.3 | 4.2 | 44.1 - 48.5 |
| | Device | 10 | 31.7 | 10.0 | 28.3 - 35.1 |
| | Overall | 34 | 42.0 | 9.2 | 38.8 - 45.3 |
| 90-101 | Male | 2 | 40.0 | 1.4 | 28.9 - 51.1 |
| | Female | 15 | 36.9 | 9.7 | 32.8 - 40.9 |
| | No Device | 7 | 45 | 4.2 | 40.9 - 49.1 |
| | Device | 10 | 31.8 | 7.6 | 28.4 - 35.2 |
| | Overall | 17 | 37.2 | 9.1 | 32.5 - 41.9 |


| Name: | Date: | |
|----------------------------------------|--------|---------|
| Location: | Rater: | |
| ITEM DESCRIPTION | SCORE | E (0-4) |
| Sitting to standing | | |
| Standing unsupported | | |
| Sitting unsupported | | |
| Standing to sitting | | |
| Transfers | | |
| Standing with eyes closed | | |
| Standing with feet together | | |
| Reaching forward with outstretched arm | | |
| Retrieving object from floor | | |
| Turning to look behind | | |
| Turning 360 degrees | | |
| Placing alternate foot on stool | | |
| Standing with one foot in front | | |
| Standing on one foot | | |
| Total | | |

### GENERAL INSTRUCTIONS

Please document each task and/or give instructions as written. When scoring, please <u>record</u> the lowest response category that applies for each item.

In most items, the subject is asked to maintain a given position for a specific time. Progressively more points are deducted if:

- · the time or distance requirements are not met
- · the subject's performance warrants supervision
- the subject touches an external support or receives assistance from the examiner Subject should understand that they must maintain their balance while attempting the tasks.
   The choices of which leg to stand on or how far to reach are left to the subject. Poor judgment will adversely influence the performance and the scoring.

Equipment required for testing is a stopwatch or watch with a second hand, and a ruler or other indicator of 2, 5, and 10 inches. Chairs used during testing should be a reasonable height. Either a step or a stool of average step height may be used for item # 12.


| ( ) 4 able to 3<br>( ) 2 able to 3<br>( ) 2 needs m | NDING Please stand up. Try not to use your hand for support. stand without using hands and stabilize independently stand independently using hands stand using hands after several tries sinimmal aid to stand or stabilize noderate or maximal assist to stand |
|---|---|
| STANDING UNST | IPPORTED. |
| | Please stand for two minutes without holding on. |
| | stand safely for 2 minutes |
| | stand 2 minutes with supervision |
| | stand 30 seconds unsupported |
| | everal tries to stand 30 seconds unsupported |
| ( )0 unable t | to stand 30 seconds unsupported |
| If a subject is able | to stand 2 minutes unsupported, score full points for sitting unsupported. Proceed to item #4. |
| SITTING WITH B | ACK UNSUPPORTED BUT FEET SUPPORTED ON FLOOR OR ON A STOOL |
| | Please sit with arms folded for 2 minutes. |
| | sit safely and securely for 2 minutes |
| | sit 2 minutes under supervision |
| ( )2 able to | able to sit 30 seconds |
| ( ) 1 able to | |
| ( )0 unable t | to sit without support 10 seconds |
| STANDING TO S | ITTING |
| INSTRUCTIONS: | |
| | ely with minimal use of hands |
| | s descent by using hands |
| | ck of legs against chair to control descent |
| | ependently but has uncontrolled descent<br>ssist to sit |
| ( ) o needs a | saist to sit |
| TRANSFERS | |
| | Arrange chair(s) for pivot transfer. Ask subject to transfer one way toward a seat with armrests and one way toward a |
| | sts. You may use two chairs (one with and one without armrests) or a bed and a chair. |
| | transfer safely with minor use of hands |
| ( )3 able to t | transfer safely definite need of hands |
| | transfer with verbal cuing and/or supervision<br>ne person to assist |
| | wo people to assist or supervise to be safe |
| ( ) 0 110011 | to people to about of supervise to be sure |
| STANDING UNST | UPPORTED WITH EYES CLOSED |
| | Please close your eyes and stand still for 10 seconds. |
| | stand 10 seconds safely |
| | stand 10 seconds with supervision |
| | stand 3 seconds |
| | to keep eyes closed 3 seconds but stays safely<br>elp to keep from falling |
| ( ) o needs n | esp to keep from failing |
| STANDING UNST | UPPORTED WITH FEET TOGETHER |
| INSTRUCTIONS: | Place your feet together and stand without holding on. |
| | place feet together independently and stand 1 minute safely |
| | place feet together independently and stand 1 minute with supervision |
| | place feet together independently but unable to hold for 30 seconds |
| | elp to attain position but able to stand 15 seconds feet together |
| ( ) 0 needs h | ein to attain notition and linante to note for ( ) seconds |


| REACHING FORWARD WITH OUTSTRETCHED ARM WHILE STANDING INSTRUCTIONS: Lift arm to 90 degrees. Stretch out your fingers and reach forward as far as you can. | |
|---|---|
| end of fingertips when arm is at 90 degrees. Fingers should not touch the ruler while reaching forward. It distance forward that the fingers reach while the subject is in the most forward lean position. When possarms when reaching to avoid rotation of the trunk.) ( ) 4 can reach forward confidently 25 cm (10 inches) | |
| ( )3 can reach forward 12 cm (5 inches)<br>( )2 can reach forward 5 cm (2 inches) | |
| ( ) 1 reaches forward but needs supervision<br>( ) 0 loses balance while trying/requires external support | |
| PICK UP OBJECT FROM THE FLOOR FROM A STANDING POSITION INSTRUCTIONS: Pick up the shoe/slipper, which is place in front of your feet. | |
| ( ) 4 able to pick up slipper safely and easily ( ) 3 able to pick up slipper but needs supervision ( ) 2 unable to pick up but reaches 2-5 cm(1-2 inches) from slipper and keeps balance | |
| independently ( ) 1 unable to pick up and needs supervision while trying | |
| ( ) 0 unable to try/needs assist to keep from losing balance or falling TURNING TO LOOK BEHIND OVER LEFT AND RIGHT SHOULDERS WHILE STANDING | |
| INSTRUCTIONS: Turn to look directly behind you over toward the left shoulder. Repeat to the right. Elook at directly behind the subject to encourage a better twist turn. ( ) 4 looks behind from both sides and weight shifts well | xaminer may pick an object to |
| looks behind one side only other side shows less weight shift turns sideways only but maintains balance | |
| ( ) 1 needs supervision when turning<br>( ) 0 needs assist to keep from losing balance or falling | |
| TURN 360 DEGREES INSTRUCTIONS: Turn completely around in a full circle. Pause. Then turn a full circle in the other dire | ection. |
| ( ) 4 able to turn 360 degrees safely in 4 seconds or less ( ) 3 able to turn 360 degrees safely one side only 4 seconds or less | |
| ( ) 2 able to turn 360 degrees safely but slowly ( ) 1 needs close supervision or verbal cuing ( ) 0 needs assistance while turning | |
| PLACE ALTERNATE FOOT ON STEP OR STOOL WHILE STANDING UNSUPPORTED INSTRUCTIONS: Place each foot alternately on the step/stool. Continue until each foot has touch the st | rep/stool four times. |
| <ul> <li>( ) 4 able to stand independently and safely and complete 8 steps in 20 seconds</li> <li>( ) 3 able to stand independently and complete 8 steps in &gt; 20 seconds</li> </ul> | |
| ( ) 2 able to complete 4 steps without aid with supervision ( ) 1 able to complete > 2 steps needs minimal assist ( ) 0 needs assistance to keep from falling/unable to try | |
| STANDING UNSUPPORTED ONE FOOT IN FRONT INSTRUCTIONS: (DEMONSTRATE TO SUBJECT) Place one foot directly in front of the other. If yo foot directly in front, try to step far enough ahead that the heel of your forward foot is ahead of the toes of | |
| points, the length of the step should exceed the length of the other foot and the width of the stance should normal stride width.) | d approximate the subject's |
| ( ) 4 able to place foot tandem independently and hold 30 seconds ( ) 3 able to place foot ahead independently and hold 30 seconds | |
| ( ) 2 able to take small step independently and hold 30 seconds ( ) 1 needs help to step but can hold 15 seconds ( ) 0 loses balance while stepping or standing | |
| STANDING ON ONE LEG INSTRUCTIONS: Stand on one leg as long as you can without holding on. | |
| ( ) 4 able to lift leg independently and hold > 10 seconds<br>( ) 3 able to lift leg independently and hold 5-10 seconds | |
| <ul> <li>( ) 2 able to lift leg independently and hold ≥ 3 seconds</li> <li>( ) 1 tries to lift leg unable to hold 3 seconds but remains standing independently.</li> <li>( ) 0 unable to try of needs assist to prevent fall</li> </ul> | |

### ( ) TOTAL SCORE (Maximum = 56)


### **Short Falls Efficacy Scale - International**

### **Short FES-I**

Now we would like to ask some questions about how concerned you are about the possibility of falling. Please reply thinking about how you usually do the activity. If you currently don't do the activity, please answer to show whether you think you would be concerned about falling IF you did the activity. For each of the following activities, please tick the box which is closest to your own opinion to show how concerned you are that you might fall if you did this activity.

| ***** | t jeu ningin ran n jeu uru tine a <b>t</b> ti | . 10) . | | | |
|---|---|---|---|---|---|
| | | Not at all | Somewhat | Fairly | Very |
| | | concerned | concerned | concerned | concerned |
| | | 1 | 2 | 3 | 4 |
| 1 | Getting dressed or undressed | 1 🗆 | 2 🗆 | 3 🗖 | 4 🗆 |
| 2 | Taking a bath or shower | 1 🗆 | 2 🗆 | 3 🗆 | 4 🗆 |
| 3 | Getting in or out of a chair | 1 🗆 | 2 🗆 | 3 🗆 | 4 🗆 |
| 4 | Going up or down stairs | 1 🗆 | 2 🗆 | 3 🗆 | 4 🗆 |
| 5 | Reaching for something above your head or on the ground | 1 🗆 | 2 🗆 | 3 🗆 | 4 🗆 |
| 6 | Walking up or down a slope | 1 🗆 | 2 🗆 | 3 🗆 | 4 🗆 |
| 7 | Going out to a social event<br>(e.g. religious service, family<br>gathering or club meeting) | 1 🗆 | 2 🗆 | 3 🗆 | 4 🗆 |

 $Kempen\ GIJM,\ Yardley\ L.,\ Haastregt\ JCM\ van,\ Zijlstra\ GAR,\ Beyer\ N,\ Hauer\ K,\ Todd\ C.$ 
